CLINICAL TRIAL: NCT00409188
Title: A Multi-center Phase III Randomized, Double-blind Placebo-controlled Study of the Cancer Vaccine Stimuvax® (L-BLP25 or BLP25 Liposome Vaccine) in Non-small Cell Lung Cancer (NSCLC) Subjects With Unresectable Stage III Disease.
Brief Title: Cancer Vaccine Study for Unresectable Stage III Non-small Cell Lung Cancer (START)
Acronym: START
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMR 63325-001
Record Dates: First submitted 2006-12-07; First posted 2006-12-08 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-Small Cell Lung Carcinoma;; stage III;; unresectable;; vaccine; Tecemotide; L-BLP25;; Cyclophosphamide;; placebo controlled;; randomized;; double blind;; immunotherapy;
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — L-BLP25; Single Person; Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tecemotide (L-BLP25) (Experimental)
  Interventions: Biological: Tecemotide (L-BLP25); Drug: Single low dose cyclophosphamide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Tecemotide (L-BLP25) — After receiving cyclophosphamide, participants will receive 8 consecutive weekly subcutaneous vaccinations with 806 microgram (mcg) of tecemotide (L-BLP25) at Weeks 0, 1, 2, 3, 4, 5, 6, and 7 followed by maintenance vaccinations with 806 mcg of tecemotide (L-BLP25) at 6-week intervals, commencing at Week 13, until disease progression is documented.
  Arms: Tecemotide (L-BLP25)
Drug: Single low dose cyclophosphamide — A single intravenous infusion of 300 milligram per square meter (mg/m^2) (to a maximum 600 mg) of cyclophosphamide will be given 3 days before first tecemotide (L-BLP25) vaccination.
  Arms: Tecemotide (L-BLP25)
Drug: Placebo — A single infusion (IV) of 0.9% Saline solution instead of cyclophosphamide but in the same calculated dose will be given three days before first placebo vaccination. Subjects will then receive eight consecutive weekly subcutaneous vaccinations with placebo at weeks 0; 1; 2; 3; 4; 5; 6 and 7 followed by maintenance placebo vaccinations at 6-week intervals, commencing at week 13, until disease progression is documented.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the cancer vaccine tecemotide (L-BLP25) in addition to best supportive care is effective in prolonging the lives of subjects with unresectable stage III non-small cell lung cancer, compared to best supportive care alone.

A local ancillary (sub) study in European centers will evaluate the immune response in peripheral blood after tecemotide (L-BLP25) or placebo vaccination.

DETAILED DESCRIPTION:
Ancillary Trial: An exploratory investigation of immune response in peripheral blood after tecemotide (L-BLP25) or placebo vaccination.

The ancillary study is a sub-study within START. This is an exploratory investigation of the immune response in peripheral blood after tecemotide (L-BLP25) or placebo vaccination. The main objective is to evaluate whether administration of single-shot, low-dose cyclophosphamide followed by tecemotide (L-BLP25) vaccinations induces specific immune response in peripheral blood to BLP25 (the mucinous glycoprotein 1 [MUC1] antigen) as well as a modulation of cellular and soluble components of the immune response in subjects with unresectable stage III NSCLC.

Twenty-five of the European START sites will participate in the ancillary study.

Sample size: up to 60 to 80 subjects

All inclusion criteria specified in the START clinical trial protocol except for hemoglobin >= 100 gram/Liter (g/L)

All exclusion criteria are the same as specified in the START clinical trial protocol

Schedule of events: Blood samples will be taken at baseline, visit week 4, 8 13 and 25 (80 milliliter (mL) whole blood each)

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented unresectable stage III non-small cell lung cancer (NSCLC)
* Documented stable disease or objective response, according to Response Evaluation Criteria in Solid Tumors (RECIST), after primary chemoradiotherapy (either sequential or concomitant) for unresectable stage III disease, within 4 weeks (28 days) prior to randomization
* Receipt of concomitant or sequential chemoradiotherapy, consisting of a minimum of two cycles of platinum-based chemotherapy and a minimum radiation dose of >=50 Gray (Gy). Subjects must have completed the primary thoracic chemo-radiotherapy at least four weeks (28 days) and no later than 12 weeks (84 days) prior to randomization. Subjects who received prophylactic brain irradiation as part of primary chemo-radiotherapy are eligible
* Geographically accessible for ongoing follow-up, and committed to comply with the designated visits
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* A platelet count > 140 x 10^9/Liter; white blood cells (WBC) > 2.5 x 10^9/Liter and hemoglobin > 90 gram per liter (g/L)

Exclusion Criteria:

Pre-Therapies:

* Undergone lung cancer specific therapy (including surgery) other than primary chemo-radiotherapy
* Receipt of immunotherapy (e.g. interferons, tumor necrosis factor [TNF], interleukins, or biological response modifiers [granulocyte macrophage colony stimulating factor {GM-CSF}, granulocyte colony stimulating factor {G-CSF}, macrophage-colony stimulating factor {M-CSF}], monoclonal antibodies) within 4 weeks (28 days) prior to randomization
* Receipt of investigational systemic drugs (including off-label use of approved products) within 4 weeks (28 days) prior to randomization

Disease Status:

* Metastatic disease
* Malignant pleural effusion at initial diagnosis and/or at study entry
* Past or current history of neoplasm other than lung carcinoma, except for curatively treated non-melanoma skin cancer, in situ carcinoma of the cervix or other cancer curatively treated and with no evidence of disease for at least 5 years
* Autoimmune disease
* A recognized immunodeficiency disease including cellular immunodeficiencies, hypogammaglobulinemia or dysgammaglobulinemia; subjects who have hereditary or congenital immunodeficiencies
* Any preexisting medical condition requiring chronic steroid or immunosuppressive therapy (steroids for the treatment of radiation pneumonitis are allowed)
* Known Hepatitis B and/or C

Physiological Functions:

* Clinically significant hepatic dysfunction
* Clinically significant renal dysfunction
* Clinically significant cardiac disease
* Splenectomy
* Infectious process that in the opinion of the investigator could compromise the subject's ability to mount an immune response

Standard Safety:

* Pregnant or breast-feeding women, women of childbearing potential, unless using effective contraception as determined by the investigator
* Known drug abuse/alcohol abuse
* Legal incapacity or limited legal capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1513 (Actual)
Dates: Start 2007-01; Primary Completion 2012-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Inc., an affiliate of Merck KGaA, Darmstadt, Germany
Locations (289):
- United States (48):
  - Saint Edward Mercy Medical Center, Fort Smith, Arkansas
  - Pacific Cancer Medical Center, Anaheim, California
  - Glendale Adventist Medical Center, Glendale, California
  - Norris Cancer Hospital, Los Angeles, California
  - Cedars-Sinai Outpatient Cancer Center at the Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - Clinical Trials and Research Associates, Inc., Montebello, California
  - Desert Hematology Oncology Medical Group, Inc, Rancho Mirage, California
  - Stockton Hematology Oncology Medical Group, Inc., Stockton, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Pasco Hernando Oncology Associates P.A, Brooksville, Florida
  - University of Miami, Sylvester Comprehensive Cancer Center, Miami, Florida
  - Pasco Hernando Oncology Associates, PA, New Port Richey, Florida
  - Florida Hospital Memorial System, Ormond Beach, Florida
  - Southern Illinois Hematology/Oncology, Centralia, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Joliet Oncology-Hematology Associates, Ltd., Joliet, Illinois
  - Kentucky Cancer Center, Hazard, Kentucky
  - Leonard J. Chabert Medical Center, Houma, Louisiana
  - Hematology and Oncology Specialists, LLC, Metarie, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - University of Maryland, Marlene and Steward Greenbaum Cancer Center, Baltimore, Maryland
  - Lahey Clinic, Burlington, Massachusetts
  - Oncology Care Associates, Saint Joseph, Michigan
  - University of Minnesota Physicians, Masonic Cancer Center, Minneapolis, Minnesota
  - Saint Louis University Cance Center, St Louis, Missouri
  - Deaconess Billings Clinic, Billings, Montana
  - Big Sky Oncology, Sletten Cancer Institute, Great Falls, Montana
  - Nebraska Cancer Care, LLC, Hastings, Nebraska
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - St. Vincents Comprehensive Cancer Center, New York, New York
  - Hematology Oncology Associates of Rockland, Nyack, New York
  - Univ. of North Carolina at Chapel Hill, Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Hematology-Oncology, Charlotte, North Carolina
  - Hanover Medical Specialts PA, Wilmington, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Signal Point Clinical Research Center, LLC, Middletown, Ohio
  - Southwestern Regional Medical Center, Tulsa, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Univ. of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - The Jones Clinic, PC, Germantown, Tennessee
  - Center for Oncology Research, Dallas, Texas
  - John Peter Smith Center for Cancer Care, Fort Worth, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Cancer Therapy & Research Center, Institute for Drug Development, San Antonio, Texas
  - Fairfax-Northern Virginia Hematology Oncology, PC, Fairfax, Virginia
  - Wheeling Hospital, Wheeling, West Virginia
- Argentina (9):
  - Hospital Italiano Regional del Sur, Bahía Blanca, Buenos Aires
  - Paliar, Capital, Buenos Aires, Buenos Aires
  - Corporacion Medica General San Martin, San Martín, Buenos Aires
  - Centro Oncologico de Roario, Rosario, Santa Fe Province
  - Centro de Educacion Medica e Investigaciones Clinicas "Norberto Quirno" (CEMIC), Buenos Aires
  - Instituto Especializado Alexander Fleming, Buenos Aires
  - Sociedad Intaliana de Beneficencia en Buenos Aires, Hospital Italiano, Buenos Aires
  - Clinica Universitaria Reina Fabiola, Córdoba
  - Research Site, Tandil
- Australia (7):
  - Research Site, Nedlands, Western Australia
  - Research Site, Bankstown, NSW
  - Research Site, Camperdown
  - Research Site, Heidelberg
  - Research Site, Kingswood
  - Research Site, Saint Leonards
  - Research Site, Woolloongabba
- Austria (7):
  - Research Site, Graz, Styria
  - Research Site, Linz, Upper Austria
  - Research Site, Inssbruck
  - Research Site, Salzburg
  - Research Site, Vienna
  - Research Site, Wein, Venna
  - Research Site, Wels
- Belgium (6):
  - Research Site, Brasschaat
  - Research Site, Brussels
  - Research Site, Haine-Saint-Paul
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Mechelen
- Brazil (15):
  - Hospital das Clinicas da Faculdade de Medinina de Univeridade, São Paulo, De Ao Paulo
  - Nugieo de Oncologia da Bahia, Salvador, Estado de Bahia
  - Hospital LifeCenter, Belo Horizonte, Minas Gerais
  - Hospital Nossa Senhora da Conceicao, Centro de Pesquisas Medicas e Ensaios Clinicos, Porto Alegre, Rio Grande Do Sol
  - Associacao Hospital de Caridade Ijui, Ijuí, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Dept. de Endocrinologia, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas-Pucrs, Porto Alegre, Rio Grande do Sul
  - Research Site, Porto Algre, Rio Grande do Sul
  - Centro de Oncologia de Campinas - OCC, Campinas, São Paulo
  - Fundacao Hospital Amaral Carvalho, Jaú, São Paulo
  - Instituto do Cancer Arnaldo Vieira de Caralho-Onco-pneumonia, São Paulo, São Paulo
  - Santa Casa de Misericordia De Sao Paulo, São Paulo, São Paulo
  - Instituto de Oncologia de Sorocaba, Sorocaba, São Paulo
  - Research Site, Ondina-Salvdor
  - Instituto Nacional do Cancer - INCA, Rio de Janeriro
- Canada (17):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Cross Cancer Institue, Edmonton, Alberta
  - Frazer Valley Cancer Center, Surrey, British Columbia
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Vancouver Island Cancer Center, Victoria, British Columbia
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Capital District Health Authority, Halifax, Nova Scotia
  - Cape Breton Districk Health Authority Cancer Care, Sydney, Nova Scotia
  - Juravinski Cancer Center, Hamilton, Ontario
  - Niagara Health System, Saint Catharines, Ontario
  - Thunder Bay Regional Health Science Center Northwestern Ontario Regional Center, Thunder Bay, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Windsor Regional Cancer Center, Windsor, Ontario
  - Hopital Notre Dame, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Hopital Laval, Sainte-Foy, Quebec
- China (3):
  - Research Site, Beijing
  - Research Site, Guangzhou
  - Research Site, Shanghai
- Czechia (4):
  - Research Site, Hradec Králové
  - Research Site, Ostrava-Poruba
  - Research Site, Prague
  - Research Site, Ústí nad Labem
- Denmark (2):
  - Research Site, Herlev
  - Research Site, Odense C
- France (13):
  - Research Site, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Research Site, Besançon, Franche-Comte
  - Research Site, Beuvry
  - Research Site, Brest
  - Research Site, Caen
  - Research Site, Chauny
  - Research Site, Marseille
  - Research Site, Nancy
  - Research Site, Nantes-Saint Herblain
  - Research Site, Paris
  - Research Site, Perpignan
  - Research Site, Poitiers
  - Research Site, Strasbourg
- Germany (24):
  - Research Site, Essen, North Rhine-Westphalia
  - Research Site, Hemer, North Rhine-Westphalia
  - Research Site, Mainz, Rhineland-Palatinate
  - Research Site, Homburg, Saarland
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Coswig
  - Research Site, Essen
  - Research Site, Frankfurt am Main
  - Research Site, Freiburg im Breisgau
  - Research Site, Gauting
  - Research Site, Großhansdorf
  - Research Site, Hamburg
  - Reseach Site, Heidelberg
  - Research Site, Kassel
  - Research Site, Kiel
  - Research Site, Leipzig
  - Research Site, Magdeburg
  - Research Site, Mainz
  - Research Site, Minden
  - Research Site, Mutzschen
  - Research Site, München
  - Research Site, Oldenburg
  - Research Site, Rostock
- Greece (6):
  - Research Site, Marousi, Athens
  - Research Site, Athens, Attica
  - Research Site, Thessaloniki, Nea Efkarpia
  - Research Site, Athens
  - Research Site, Chidari, Athens
  - Research Site, Heraklion
- Hong Kong (2):
  - Research Site, Shatin, New Territories
  - Research Site, Hong Kong
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Mátraháza
  - Research Site, Nyíregyháza
  - Research Site, Tatabayana
- India (5):
  - Research Site, Chennai
  - Research Site, Hyderabad
  - Research Site, Mumbai
  - Research Site, New Delhi
  - Research Site, Vellore
- Research Site, Dublin, Ireland
- Israel (8):
  - Research Site, Tel Litwinsky, Tel Avir
  - Research Site, Beersheba
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Tel Aviv
  - Research Site, Ẕerifin
- Italy (17):
  - Research Site, Genova, Genova
  - Research Site, Palermo, Palermo
  - Research Site, Candiolo, Torino
  - Research Site, Avelino
  - Research Site, Bologna
  - Research Site, Carpi
  - Research Site, Chieti
  - Research Site, Forlì
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Orbassano-Torino
  - Research Site, Parma
  - Research Site, Rome
  - Research Site, Rozzano-Milano
  - Research Site, Sassari
  - Research Site, Trento
- Mexico (3):
  - Centro Oncologico de Chihuahua, Chihuahua City, Chihuahua
  - Consultorio del, Morelia, Michoacán
  - Instituto Nacional de Cancerologia (INCAN), Mexico City
- Netherlands (6):
  - Research Site, Amsterdam, North Holland
  - Research Site, Amsterdam
  - Research Site, Eindhoven
  - Research Site, Hoofdrop
  - Research Site, Tilburg
  - Research Site, Zwolle
- Poland (15):
  - Research Site, Warsaw, Masovian Voivodeship
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Bytom
  - Research Site, Gdynia
  - Research Site, Krakow
  - Genova, Lodz
  - Research Site, Olsztyn
  - Research Site, Otwock
  - Research Site, Poznan
  - Research Site, Torun
  - Genova, Warsaw
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Zabrze
- Portugal (4):
  - Genova, Coimbra
  - Genova, Lisbon
  - Genova, Porto
  - Genova, Santa Maria de Feira
- Romania (6):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Iași
  - Research Site, Sibiu
  - Research Site, Suceava
  - Research Site, Timișoara
- Russia (11):
  - Reseaerch Site, Kazan', Tatarstan Republic
  - Research Site, Yaroslavl, Yaroslavlr
  - Research Site, Barnaul
  - Genova, Chelaybinsk
  - Research Site, Ivanovo
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Obninsk
  - Research Site, Saint Petersburg
  - Research Site, Tomsk
  - Research Site, Voronezh
- Research Site, Singapore, Singapore
- Slovakia (3):
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Nitra
- South Korea (3):
  - Research Site, Goyang-si, Gyeonggi-do
  - Research Site, Seoul, Gyeonggi-do
  - Research Site, Seoul
- Spain (12):
  - Research Site, Mataró, Barcelona
  - Research Site, Barakaldo, Bilbao
  - Research Site, Donostia / San Sebastian, Guipuzcoa
  - Research Site, Jaén, Jaen
  - Research Site, A Coruña
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, Burgos
  - Research Site, Girona
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Málaga
- Sweden (6):
  - Research Site, Gävle
  - Research Site, Gothenburg
  - Research Site, Lund
  - Research Site, Stockholm
  - Research Site, Umeå
  - Research Site, Uppsala
- Switzerland (3):
  - Research Site, Basel
  - Research Site, Geneva
  - Research Site, Winterthur
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- United Kingdom (13):
  - Research Site, Cornwall
  - Research Site, Edinburgh
  - Research Site, Glasgow
  - Research Site, Guildford
  - Research Site, Inverness
  - Research Site, Leeds
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Metropolitan Borough of Wirral
  - Research Site, Southampton
  - Research Site, Surrey
  - Research Site, Torquay

REFERENCES:
- [Background] Butts C, Socinski MA, Mitchell P, Thatcher N, Havel L, Krzakowski M, Nawrocki S, Ciuleanu TE, Bosquée L, Trigo JM, Spira A, Tremblay L, Nyman J, Ramlau R, Helwig C, Falk MH, Shepherd FA. START: A phase III study of L-BLP25 cancer immunotherapy for unresectable stage III non-small cell lung cancer. American Society of Clinical Oncology - 49th Annual Meeting. 2013; Abstr No. 7500.
- [Background] Shepherd FA, Socinski MA, Mitchell P, Thatcher N, Havel L, Krzakowski M, Nawrocki S, Helwig C, Schroeder A, Butts C. Updated analysis and secondary endpoints with L-BLP25 in unresectable stage III non-small cell lung cancer in the phase III START study. European Society for Medical Oncology 38th Congress - ECCO 17, ESMO 38, ESTRO 32. 2013. Abstr No. 3419.
- [Background] Mitchell P, Butts C, Socinski M, Thatcher N, Wichardt-Johansson G, Ellis P, Gladkov O, Pereira J, Eberhardt W, Horwood K, Szczesna A, Helwig C, Schröder A, Shepherd F. Tecemotide (L-BLP25) in unresectable stage III non-small cell lung cancer in the phase III START study: Further endpoint and exploratory biomarker results. World Conference on Lung Cancer - 15th. 2013; Abstr. No. 2779.
- [Background] Thatcher N, Shepherd FA, Mitchell P, Socinski MA, Paredes A, Lambrechts M, Thomas M, Kollmeier J, Zemanová M, Sadjadian P, Peylan-Ramu N, Helwig C, Schröder A, Butts C. Geographic differences in the combined-modality treatment of stage III unresectable non-small cell lung cancer: Results from a global phase III trial of tecemotide (L-BLP25). World Conference on Lung Cancer - 15th. 2013; Abstr. No. 2712.
- [Background] Socinski M, Butts C, Mitchell P, Thatcher N, Scagliotti G, Robinet G, Martin C, Zukin M, Ragulin Y, Bonomi P, Yang CH, Regnault A, Helwig C, de Nigris E, Shepherd F. Exploration of patient health status as measured by the generic preference-based questionnaire EQ-5D alongside the START trial of tecemotide in non-small cell lung cancer. World Conference on Lung Cancer - 15th. 2013; Abstr. No. 2744.
- [Result] Butts C, Socinski MA, Mitchell PL, Thatcher N, Havel L, Krzakowski M, Nawrocki S, Ciuleanu TE, Bosquee L, Trigo JM, Spira A, Tremblay L, Nyman J, Ramlau R, Wickart-Johansson G, Ellis P, Gladkov O, Pereira JR, Eberhardt WE, Helwig C, Schroder A, Shepherd FA; START trial team. Tecemotide (L-BLP25) versus placebo after chemoradiotherapy for stage III non-small-cell lung cancer (START): a randomised, double-blind, phase 3 trial. Lancet Oncol. 2014 Jan;15(1):59-68. doi: 10.1016/S1470-2045(13)70510-2. Epub 2013 Dec 9. PMID 24331154
- [Result] DeGregorio M, Soe L, Wolf M. Tecemotide (L-BLP25) versus placebo after chemoradiotherapy for stage III non-small cell lung cancer (START): a randomized, double-blind, phase III trial. J Thorac Dis. 2014 Jun;6(6):571-3. doi: 10.3978/j.issn.2072-1439.2014.05.15. No abstract available. PMID 24976972
- [Derived] Zhu J, Yuan Y, Wan X, Yin D, Li R, Chen W, Suo C, Song H. Immunotherapy (excluding checkpoint inhibitors) for stage I to III non-small cell lung cancer treated with surgery or radiotherapy with curative intent. Cochrane Database Syst Rev. 2021 Dec 6;12(12):CD011300. doi: 10.1002/14651858.CD011300.pub3. PMID 34870327
- [Derived] Mitchell P, Thatcher N, Socinski MA, Wasilewska-Tesluk E, Horwood K, Szczesna A, Martin C, Ragulin Y, Zukin M, Helwig C, Falk M, Butts C, Shepherd FA. Tecemotide in unresectable stage III non-small-cell lung cancer in the phase III START study: updated overall survival and biomarker analyses. Ann Oncol. 2015 Jun;26(6):1134-1142. doi: 10.1093/annonc/mdv104. Epub 2015 Feb 26. PMID 25722382

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last participant (informed consent): 25 January 2007/31 October 2011. Data cut-off for primary endpoint analysis: 08 August 2012. Participants randomized at 264 centers in 33 countries worldwide.
Pre-assignment Details: A total of 1908 participants were screened for eligibility and 1513 participants were enrolled and randomized.
Groups:
- Tecemotide (L-BLP25) + Cyclophosphamide: A single intravenous infusion of 300 milligram per square meter (mg/m^2) (to a maximum 600 mg) of cyclophosphamide was given 3 days before first tecemotide (L-BLP25) vaccination. After receiving cyclophosphamide, participants received 8 consecutive weekly subcutaneous vaccinations with 806 microgram (mcg) of tecemotide (L-BLP25) at Weeks 0, 1, 2, 3, 4, 5, 6, and 7 followed by maintenance vaccinations with 806 mcg of tecemotide (L-BLP25) at 6-week intervals, commencing at Week 13, until disease progression was documented.
- Saline + Placebo: A single intravenous infusion of 0.9 percent (%) saline solution in the same calculated dose as cyclophosphamide was given 3 days before first placebo vaccination. After receiving saline, participants received 8 consecutive weekly subcutaneous vaccinations with placebo at Weeks 0, 1, 2, 3, 4, 5, 6, and 7 followed by maintenance placebo vaccinations at 6-week intervals, commencing at Week 13, until disease progression was documented.
Period: Overall Study
Arm/Group | Tecemotide (L-BLP25) + Cyclophosphamide | Saline + Placebo
Started | 1006 | 507
Completed | 623 | 332
Not Completed | 383 | 175
Not completed — Ongoing at data cut-off | 383 | 175

BASELINE CHARACTERISTICS:
Population: ITT population included all the subject who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tecemotide (L-BLP25) + Cyclophosphamide | Saline + Placebo | Total
Number analyzed (Participants) | 1006 | 507 | 1513
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (9.1) | 60.9 (9.0) | 60.8 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 315 | 162 | 477
  Male | 691 | 345 | 1036

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival time was defined as the time from randomization to death. Participants without events were censored at the last date they were known to be alive or the clinical cut-off date, whatever was earlier.
Time Frame: Up to 66 months
Population: Primary analysis set (modified intention-to-treat [ITT] population) was based on the ITT population but prospectively excluded all participants (274 participants) that were randomized during the 6 months (22 Sep 2009 to 22 Mar 2010) prior to the effective date of clinical hold.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tecemotide (L-BLP25) + Cyclophosphamide | Saline + Placebo
Number analyzed (Participants) | 829 | 410
months | 25.6 [22.5 to 29.2] | 22.3 [19.6 to 25.5]
Statistical Analysis 1: Comparison: Tecemotide (L-BLP25) + Cyclophosphamide vs Saline + Placebo; Test type: Superiority or Other; p = 0.1566, Regression, Cox; Hazard Ratio (HR) = 0.893, 95% CI 2-sided [0.763 to 1.044]

2. Secondary Outcome: Time To Symptom Progression (TTSP) as Measured by the Lung Cancer Symptom Scale (LCSS)
Description: Time to symptom progression (TTSP) was measured by LCSS. Symptomatic progression was defined as an increase (worsening) of the Average Symptomatic Burden Index (ASBI that is, the mean of the six major lung cancer specific symptom scores of the LCSS patient scale - ranging from 0 to 100 where higher score indicates worst outcome). Worsening was defined as a 10% increase in the scale breadth from the baseline score. TTSP is defined as the time from randomization to worsening in ASBI. Participants without event are censored at the date of the last LCSS assessment.
Time Frame: Up to 66 months
Population: Primary analysis set (modified ITT population) was based on the ITT population but prospectively excluded all participants (274 participants) that were randomized during the 6 months (22 Sep 2009 to 22 Mar 2010) prior to the effective date of clinical hold. "N" signifies the number of participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tecemotide (L-BLP25) + Cyclophosphamide | Saline + Placebo
Number analyzed (Participants) | 829 | 409
months | 14.2 [12.9 to 15.7] | 11.4 [9.3 to 13.1]
Statistical Analysis 1: Comparison: Tecemotide (L-BLP25) + Cyclophosphamide vs Saline + Placebo; Test type: Superiority or Other; p = 0.0226, Regression, Cox; Hazard Ratio (HR) = 0.845, 95% CI 2-sided [0.732 to 0.977]

3. Secondary Outcome: Time To Progression (TTP)
Description: Time from randomization to disease progression. Disease progression was defined based on Response Evaluation Criteria in Solid Tumors Version 1.0 [RECIST v1.0]) as at least a 20% increase in the sum of the longest diameter of target lesions from nadir, or the appearance of one or more new lesions.
Time Frame: Up to 66 months
Population: Primary analysis set (modified ITT population) was based on the ITT population but prospectively excluded all participants (274 participants) that were randomized during the 6 months (22 Sep 2009 to 22 Mar 2010) prior to the effective date of clinical hold.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tecemotide (L-BLP25) + Cyclophosphamide | Saline + Placebo
Number analyzed (Participants) | 829 | 410
months | 10.0 [9.1 to 11.5] | 8.4 [7.2 to 10.8]
Statistical Analysis 1: Comparison: Tecemotide (L-BLP25) + Cyclophosphamide vs Saline + Placebo; Test type: Superiority or Other; p = 0.0528, Regression, Cox; Hazard Ratio (HR) = 0.868, 95% CI 2-sided [0.752 to 1.002]

4. Secondary Outcome: One-, Two- and Three-year Survival Rate
Description: The percentages of participants who were alive at 1, 2, and 3 years were calculated as a cumulative percentage by Kaplan-Meier survival analysis approach.
Time Frame: Years 1, 2, and 3
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Tecemotide (L-BLP25) + Cyclophosphamide | Saline + Placebo
Number analyzed (Participants) | 829 | 410
percentage of participants
  Year 1 | 77.0 | 74.7
  Year 2 | 50.8 | 45.9
  Year 3 | 40.2 | 37.0

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events and Injection Site Reactions
Description: Treatment -emergent adverse events were defined as those with onset or worsening occurring at or after the first dosing day of study medication and up to 42 days after the last administration of any study drug or the clinical cut-off date. Injection site reactions were reported as assessed by the Investigator.
Time Frame: From first dose up to 42 days after the last dose of the trial treatment
Population: Safety analysis set included all participants who received at least 1 dose of trial treatment (cyclophosphamide, tecemotide, saline, or placebo). Participants were reported based on the actual treatment received (as-treated).
Measure: Number; unit: participants
Arm/Group | Tecemotide (L-BLP25) + Cyclophosphamide | Saline + Placebo
Number analyzed (Participants) | 1024 | 477
participants
  Treatment Emergent Adverse events | 938 | 432
  Injection site reaction | 176 | 56

ADVERSE EVENTS:
Time Frame: Up to 66 months
Description: Safety analysis set included all participants who received at least 1 dose of trial treatment (cyclophosphamide, tecemotide, saline, or placebo). Participants were reported based on the actual treatment received (as-treated).
Arm/Group | Tecemotide (L-BLP25) + Cyclophosphamide | Saline + Placebo
Serious Adverse Events (participants affected / at risk) | 303/1024 | 151/477
Other Adverse Events (participants affected / at risk) | 918/1024 | 417/477
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tecemotide (L-BLP25) + Cyclophosphamide (N=1024) | Saline + Placebo (N=477)
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Hypocoagulable state (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 3 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 4
Angina pectoris (Cardiac disorders) | 3 | 3
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 8 | 3
Atrial flutter (Cardiac disorders) | 3 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 2 | 2
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 3 | 1
Myocardial ischaemia (Cardiac disorders) | 2 | 0
Palpitations (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 3 | 1
Pericarditis (Cardiac disorders) | 2 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 2 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 2
Adrenal insufficiency (Endocrine disorders) | 2 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Retinal vascular thrombosis (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Aphagia (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 4 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Hernial eventration (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 2
Intestinal infarction (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal dilatation (Gastrointestinal disorders) | 1 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 2 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3
Asthenia (General disorders) | 2 | 3
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 9 | 3
Death (General disorders) | 2 | 0
Disease progression (General disorders) | 6 | 11
Fatigue (General disorders) | 3 | 0
Gait disturbance (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 2 | 3
Malaise (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 4 | 1
Pain (General disorders) | 1 | 1
Performance status decreased (General disorders) | 0 | 1
Pyrexia (General disorders) | 8 | 0
Spinal pain (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 4 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Helicobacter gastritis (Infections and infestations) | 1 | 0
Herpes zoster disseminated (Infections and infestations) | 1 | 0
Infectious pleural effusion (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 9 | 4
Lung abscess (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 4 | 0
Mastitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Pleural infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 30 | 14
Pneumonia primary atypical (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 7 | 2
Salmonella sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Radiation associated pain (Injury, poisoning and procedural complications) | 1 | 0
Radiation myelopathy (Injury, poisoning and procedural complications) | 0 | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 7 | 5
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic lung injury (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Wound evisceration (Injury, poisoning and procedural complications) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 32 | 9
Metastases to kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Metastases to large intestine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to small intestine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 1
Balance disorder (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 1 | 0
Carotid artery dissection (Nervous system disorders) | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 1 | 0
Cataplexy (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Convulsion (Nervous system disorders) | 4 | 2
Dizziness (Nervous system disorders) | 4 | 0
Epilepsy (Nervous system disorders) | 2 | 2
Grand mal convulsion (Nervous system disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 0
Hemiparesis (Nervous system disorders) | 4 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 1
Monoparesis (Nervous system disorders) | 1 | 0
Nerve root compression (Nervous system disorders) | 1 | 0
Paraplegia (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 1
Status epilepticus (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 4 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 3 | 1
Depression (Psychiatric disorders) | 1 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Spermatocele (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29 | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 11 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Laryngeal cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 13 | 12
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 | 2
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Pericardial drainage (Surgical and medical procedures) | 1 | 0
Aortic aneurysm (Vascular disorders) | 5 | 1
Aortic stenosis (Vascular disorders) | 0 | 1
Arterial occlusive disease (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Embolism (Vascular disorders) | 1 | 0
Femoral arterial stenosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Temporal arteritis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tecemotide (L-BLP25) + Cyclophosphamide (N=1024) | Saline + Placebo (N=477)
Constipation (Gastrointestinal disorders) | 75 | 26
Diarrhoea (Gastrointestinal disorders) | 85 | 46
Nausea (Gastrointestinal disorders) | 140 | 39
Vomiting (Gastrointestinal disorders) | 65 | 26
Asthenia (General disorders) | 71 | 29
Chest pain (General disorders) | 130 | 43
Fatigue (General disorders) | 195 | 102
Influenza like illness (General disorders) | 45 | 27
Non-cardiac chest pain (General disorders) | 57 | 24
Pyrexia (General disorders) | 80 | 41
Bronchitis (Infections and infestations) | 83 | 38
Nasopharyngitis (Infections and infestations) | 128 | 44
Upper respiratory tract infection (Infections and infestations) | 96 | 37
Radiation pneumonitis (Injury, poisoning and procedural complications) | 77 | 30
Decreased appetite (Metabolism and nutrition disorders) | 109 | 44
Arthralgia (Musculoskeletal and connective tissue disorders) | 108 | 33
Back pain (Musculoskeletal and connective tissue disorders) | 146 | 52
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 54 | 22
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 92 | 33
Myalgia (Musculoskeletal and connective tissue disorders) | 73 | 18
Pain in extremity (Musculoskeletal and connective tissue disorders) | 69 | 29
Dizziness (Nervous system disorders) | 87 | 37
Headache (Nervous system disorders) | 123 | 54
Insomnia (Psychiatric disorders) | 64 | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 336 | 133
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 225 | 103
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 60 | 32
Rash (Skin and subcutaneous tissue disorders) | 53 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study, an integrated clinical and statistical study report shall be written by the Sponsor in consultation with the Coordinating Investigator based on the protocol. The first publication will be a full publication of all data from all sites. The Sponsor is entitled to delay publication in order to obtain patent protection. The ICMJE criteria for authorship will be followed. A separate publication plan will be set up to describe further publications.